CLINICAL TRIAL: NCT01119014
Title: Tolerance and Effect of Antipsychotics in Children and Adolescents With Psychosis- An Investigator-initiated, Phase IV, Randomised Double-blind Multi-centre Trial of the Benefits and Harms of Aripiprazole Versus Quetiapine in Children and Adolescents With Psychosis
Brief Title: Tolerance and Effect of Antipsychotics in Children and Adolescents With Psychosis
Acronym: TEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anne Katrine Pagsberg (Other)
Collaborators: The Psychiatric Centre for Children and Adolescents in Bispebjerg, Denmark (Unknown); Psychiatric Centre Copenhagen, Denmark (Unknown); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Albert Einstein College of Medicine (Other); Research Institute for Biological Psychiatry, Sct. Hans Hospital, Denmark (Unknown); Capital Region Pharmacy, Denmark (Unknown); The Research Council for Health and Disease, Denmark (Other); Allocated inheritance from Elizabeth Stevn and Niels Rindom, Denmark (Unknown); AP Moeller Foundation (Other); Tryg Fonden, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Anne Katrine Pagsberg, MD., PhD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEAprotocolversion5-11 03 2010; 2009-016715-38 (EudraCT Number)
Record Dates: First submitted 2010-05-03; First posted 2010-05-07 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Psychosis
Keywords: Aripiprazole; Quetiapine; Psychosis; Child; Adolescent
MeSH Terms: conditions — Psychotic Disorders | interventions — Aripiprazole; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripirazole (Experimental)
  Interventions: Drug: Aripiprazole
- Quetiapine prolong (Experimental)
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Aripiprazole — pill, 2,5-20 mg/day, maximum 16 weeks
  Arms: Aripirazole
Drug: Quetiapine — pill, 50-600mg/day, maximum 16 weeks
  Arms: Quetiapine prolong

SUMMARY:
The benefits and harms of antipsychotics are relatively well studied in adults. However, there is a lack of scientifically valid studies regarding the benefits and harms of antipsychotics in children and adolescents with psychosis.

The main objective of the TEA trial is to compare the efficacy and adverse reactions of two antipsychotics (quetiapine versus aripiprazole) in children and adolescents between 12-17 years of age with psychotic symptoms on psychopathology, cognitive deficits, and daily functioning. Furthermore, the trial will focus on adverse reaction profiles of the two antipsychotics as well as early predictors of later sustained clinical effects of these antipsychotics.

DETAILED DESCRIPTION:
A sex and age matched healthy control group will be included to form a reference group for cognitive and somatic measures. The healthy controls will not receive any trial medication.

ELIGIBILITY:
Patients - Inclusion Criteria:

* Diagnosis: Children and adolescents with a non-organic and non-drug-induced psychosis, meeting the criteria for ICD-10 diagnoses: F20, F22-F29 and F30.2, F31.2 F31.5, F32.3 and F33.3. This is verified with a semi-structured psychopathological interview using K-SADS-PL (Kaufmann 1997) four weeks after inclusion into the trial.
* Psychopathology: Children and adolescents with psychotic symptoms, scoring ≥ 4 on at least one of the following PANSS items: P1 (delusions), P2 (conceptual disorganisation), P3 (hallucinations), P5 (grandiosity), P6 (suspiciousness/persecution) or G9 (unusual thought content); and a total PANSS score > 60. The treating physician has decided to prescribe an antipsychotic compound.
* Age: 12-17 years (both inclusive).
* Sex: Both sexes are included.
* Previous treatment: Patients must be antipsychotic-naïve. The maximum accepted previous treatment with antipsychotic compounds is two weeks cumulatively, and during the two weeks prior to inclusion no continuous treatment and a maximum of four dosages in total can have been received.
* Somatic illness: No somatic contraindication to planned medication, documented by standard somatic examination
* Written informed consent.

Patients - Exclusion Criteria:

* Compulsory treatment: Patients that are compulsorily hospitalised against their will are excluded. If their status changes to voluntary hospitalisation, patients can be included. If the patient is already included in the trial and is briefly detained, confined, or subjected to other forceful treatment according to the Danish Psychiatric Care Act ('Psykiatriloven'), both the patient and parents have to agree to remain in the trial if exclusion is to be avoided. Compulsory treatment in the form of, e.g., brief forced immobilisation or single instances of forced medication, are not causes for exclusion.
* Diagnoses: Patients with drug-induced or organic psychosis, severe chronic somatic illness, or a history of severe head-trauma are not included. Patients that do not have psychotic symptoms but are prescribed antipsychotic treatment on the indication of, e.g., severe behavioural problems or tics are not included.
* Pregnancy: Pregnant or lactating patients are not included (a pregnancy test is undertaken at inclusion). Female participants, that are sexually active, must use safe contraception throughout the trial period (see section 6.4)
* Substance abuse: People with severe alcohol or drug abuse are not included. Possible abuse is monitored both by interviewing participants and by taking a urine sample at inclusion and at 4, 12 and 52 weeks follow-up (if there is suspicion of substance abuse), testing for the presence of cocaine, amphetamine, cannabis, opiates, metamfetamine (inclusive for extacy), and benzodiazepines. When severe abuse is suspected during the trial, an ad hoc urine sample is taken. Brief periods of large alcohol/cannabis intake are not a cause of exclusion from the trial; however, cognitive and other examinations are not carried out while patients are under the influence of drugs or alcohol.
* Aggravation: Patients may be excluded if there is a significant worsening of clinical state during the course of the trial (i.e., increases of 30% or more from baseline on the PANSS total score).
* Allergy and intolerance: Patients with allergy towards the investigational drugs, or is lactose intolerant are not included.
* Lack of informed consent.

Healthy volunteers - Inclusion Criteria:

* Matching: Healthy controls (n=100) are included, in the way that they are matched to the first 100 patients included in the study (i.e., corresponding to the number of patients required in each treatment group). They will be matched according to:

  * age;
  * sex; and
  * socioeconomic status (based on a combination of parental education and income, according to criteria from the National Institute of Public Health (earlier Danish Institute of Clinical Epidemiology, DIKE)).
* Informed consent.

Healthy volunteers - Exclusion Criteria:

* Psychopathology: People with a previous psychotic disorder (ICD 10, F20-F29 and F30.2, F31.2, F31.5, F32.3 and F33.3) or current psychiatric disorder (multiaxial axis 1) are not included. This is verified by diagnostic screening using K-SADS-PL at eligibility assessment before inclusion into the study of healthy controls. The presence of psychotic psychiatric diagnoses in first-degree relatives is also a cause for exclusion.
* Somatic illnesses: People with severe chronic somatic illness or a history of severe head-trauma are not included.
* Intelligence: People with known mild mental retardation (i.e., IQ between 50-70) prior to inclusion are excluded; however, if mild mental retardation is found during the study, participants are not excluded, since they must be considered a marginal part of the normal distribution. People with moderate to severe mental retardation (i.e., IQ < 50) are excluded.
* Substance abuse: People with severe alcohol- or drug abuse are excluded. Possible abuse is monitored both by interviewing participants and by taking a urine sample at inclusion and at 4, 12 and 52 weeks follow-up (if there is suspicion of substance abuse), testing for the presence of cocaine, amphetamine, cannabis, opiates, metamfetamine (inclusive for extacy) and benzodiazepines. Brief periods of large alcohol/cannabis intake are not a cause of exclusion from the study; however, cognitive and other examinations are not carried out while participants are under the influence.
* Lack of informed consent.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2010-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Psychopathology: improvement on PANSS positive scale (PANSS 'Positive and Negative Syndrome Scale') | 12 weeks

SECONDARY OUTCOMES:
Psychopathology | 12 weeks
  Psychopathology (other PANSS scales, DIPI, SGI-S, CGI-I,and GAPD).
Cognition | 12 weeks
  Cognition and functioning (BACS Global Score, SCoRS-DK, Schizophrenia Cognition Rating Scale, BRIEF)
Adverse reactions | 12 weeks
  Adverse reactions (UKU side effect scale, AIMS, SAS, BARS, and other adverse events)
Suicidal ideation | 12 weeks
  Suicidal ideation (K-SADS-PL, specific questions for depressive disorders (current)
Genetic and antipsychotic laboratory tests | 12 weeks
  Genetic variants affecting metabolism of antipsychotics
Prognostic factors | 12 weeks
  Prognostic factors (DUP, and PAS)
Quality of Life | 52 weeks
  Quality of Life (measured with Kidscreen)
Stigmatization | 52 weeks
  Qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Anne Katrine Pagsberg, MD, Ph.D., Principal Investigator — Bispebjerg Centre for Child and Adolescent Psychiatry. University of Copenhagen.; Pia Jeppesen, MD, Ph.D., Principal Investigator — Glostrup Centre for Child and Adolescent Psychiatry. University of Copenhagen.; Maj-Britt Lauritsen, MD, Principal Investigator — Hillerød Centre for Child and Adolescent Psychiatry.; Per Hove-Thomsen, Professor, MD, D.M.Sci., Principal Investigator — Psychiatric Hospital for Children and Adolescents, Aarhus University Hospital.; Marlene Briciet Lauritsen, MD., Principal Investigator — Child- and Adolescent Psychiatric Department, Aalborg.; Niels Bilenberg, Professor, MD., Principal Investigator — Child and Adolescent Psychiatric Department, University of Southern Denmark, Odense; Thomas Werge, Professor, Ph.D., Principal Investigator — Research Institute for Biological Psychiatry, Sct. Hans Hospital, Roskilde.; Anders Fink-Jensen, MD, professor, DMSci., Principal Investigator — Psychiatric Centre Copenhagen. University of Copenhagen.; Jesper Pedersen, MD., Principal Investigator — Psychiatric Hospital for Children and Adolescent; Region Zeeland
Locations (9):
- Denmark (9):
  - Aalborg Psychiatric Hospital, Aalborg
  - Psychiatric Centre Copenhagen, Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Glostrup Hospital, Glostrup Municipality
  - Hillerød Hospital, Hillerød
  - Odense University Hospital, Odense
  - Psychiatric Hospital for Children and Adolescents, Aarhus, Risskov
  - Child and Adolescent Psychiatric Department, Region Zealand, Roskilde
  - Psychiatric Centre Sct. Hans, Roskilde

REFERENCES:
- [Derived] Klauber DG, Christensen SH, Fink-Jensen A, Pagsberg AK. I Didn't Want the Psychotic Thing to Get Out to Anyone at All: Adolescents with Early Onset Psychosis Managing Stigma. Cult Med Psychiatry. 2024 Sep;48(3):569-590. doi: 10.1007/s11013-024-09859-3. Epub 2024 Jun 13. PMID 38869653
- [Derived] Pagsberg AK, Krogmann A, Jeppesen P, von Hardenberg L, Klauber DG, Jensen KG, Ruda D, Decara MS, Jepsen JRM, Fagerlund B, Fink-Jensen A, Correll CU, Galling B. Early Antipsychotic Nonresponse as a Predictor of Nonresponse and Nonremission in Adolescents With Psychosis Treated With Aripiprazole or Quetiapine: Results From the TEA Trial. J Am Acad Child Adolesc Psychiatry. 2022 Aug;61(8):997-1009. doi: 10.1016/j.jaac.2021.11.032. Epub 2022 Jan 10. PMID 35026408
- [Derived] Jensen KG, Correll CU, Ruda D, Klauber DG, Decara MS, Fagerlund B, Jepsen JRM, Eriksson F, Fink-Jensen A, Pagsberg AK. Cardiometabolic Adverse Effects and Its Predictors in Children and Adolescents With First-Episode Psychosis During Treatment With Quetiapine-Extended Release Versus Aripiprazole: 12-Week Results From the Tolerance and Effect of Antipsychotics in Children and Adolescents With Psychosis (TEA) Trial. J Am Acad Child Adolesc Psychiatry. 2019 Nov;58(11):1062-1078. doi: 10.1016/j.jaac.2019.01.015. Epub 2019 Mar 9. PMID 30858012
- [Derived] Jensen KG, Gartner S, Correll CU, Ruda D, Klauber DG, Stentebjerg-Olesen M, Fagerlund B, Jepsen JR, Fink-Jensen A, Juul K, Pagsberg AK. Change and dispersion of QT interval during treatment with quetiapine extended release versus aripiprazole in children and adolescents with first-episode psychosis: results from the TEA trial. Psychopharmacology (Berl). 2018 Mar;235(3):681-693. doi: 10.1007/s00213-017-4784-5. Epub 2017 Nov 29. PMID 29185022
- [Derived] Pagsberg AK, Jeppesen P, Klauber DG, Jensen KG, Ruda D, Stentebjerg-Olesen M, Jantzen P, Rasmussen S, Saldeen EA, Lauritsen MG, Bilenberg N, Stenstrom AD, Nyvang L, Madsen S, Werge TM, Lange T, Gluud C, Skoog M, Winkel P, Jepsen JRM, Fagerlund B, Correll CU, Fink-Jensen A. Quetiapine extended release versus aripiprazole in children and adolescents with first-episode psychosis: the multicentre, double-blind, randomised tolerability and efficacy of antipsychotics (TEA) trial. Lancet Psychiatry. 2017 Aug;4(8):605-618. doi: 10.1016/S2215-0366(17)30166-9. Epub 2017 Jun 7. PMID 28599949
- [Derived] Jensen KG, Correll CU, Ruda D, Klauber DG, Stentebjerg-Olesen M, Fagerlund B, Jepsen JRM, Fink-Jensen A, Pagsberg AK. Pretreatment Cardiometabolic Status in Youth With Early-Onset Psychosis: Baseline Results From the TEA Trial. J Clin Psychiatry. 2017 Sep/Oct;78(8):e1035-e1046. doi: 10.4088/JCP.15m10479. PMID 28102978
- [Derived] Pagsberg AK, Jeppesen P, Klauber DG, Jensen KG, Ruda D, Stentebjerg-Olesen M, Jantzen P, Rasmussen S, Saldeen EA, Lauritsen MB, Bilenberg N, Stenstrom AD, Pedersen J, Nyvang L, Madsen S, Lauritsen MB, Vernal DL, Thomsen PH, Paludan J, Werge TM, Winge K, Juul K, Gluud C, Skoog M, Wetterslev J, Jepsen JR, Correll CU, Fink-Jensen A, Fagerlund B. Quetiapine versus aripiprazole in children and adolescents with psychosis--protocol for the randomised, blinded clinical Tolerability and Efficacy of Antipsychotics (TEA) trial. BMC Psychiatry. 2014 Jul 11;14:199. doi: 10.1186/1471-244X-14-199. PMID 25015535